CLINICAL TRIAL: NCT03597880
Title: Evaluation of Airway on Undervent Bariatric Surgery Patients
Brief Title: Preoperative Evaluation of Airway
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University Hospital (Other)
Responsible Party: Principal Investigator, nurcan kizilcik, Assist.Prof.Dr., Yeditepe University Hospital
Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: YeditepeUH
Record Dates: First submitted 2018-05-16; First posted 2018-07-24 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Obesity; Difficult Intubation
Keywords: difficult airway, obese patient,
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: retrospective clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- obese patient (Other): BMI>30 kg/m2 and underwent bariatric surgery
  Interventions: Other: obese patients

INTERVENTIONS:
Other: obese patients — underwent bariatric surgery

SUMMARY:
Evaluation of airway markers of patients who have undergone obesity surgery.

DETAILED DESCRIPTION:
The investigators evaluated the airway parameters recorded preoperatively for patients with BMI> 30 who were undervent bariatric surgery between 2015-2018 in terms of difficult airway.

ELIGIBILITY:
Inclusion Criteria:

1. BMI>30kg/m2
2. 18<age <65
3. elective surgery planned
4. ASA II-III

Exclusion Criteria:

1. BMI<30kg/m2
2. 18>age >65
3. ASA IV

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 489 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
airway evaluation for menagement in obese patient | 3 year
  preoperative airway measurements routinely performed (mallampati score, thyromental distance, neck circumference ..)for each patient will be evaluated
mallampati score | 3 year
  Class I : Visualization of the soft palate, fauces; uvula, anterior and the posterior pillars. Class II : Visualization of the soft palate, fauces and uvula. Class III : Visualization of soft palate and base of uvula. Class IV: Only hard palate is visible. Soft palate is not visible at all.
thyromental distance | 3 year
  TMD was measured as straight distance between thyroid notch and lower border of mental prominence.(cm)
neck circumference | 3 year
  Neck Circumference was measured in the midway of the neck, between mid-cervical spine and mid anterior neck, to within 1 mm, using non-stretchable plastic tape with the subjects standing upright.

CONTACTS AND LOCATIONS:
Overall Officials: nurcan kizilcik, Principal Investigator — Yeditepe UH

IPD SHARING:
Plan to Share IPD: Yes
For the protection of personal data, was decided that the personal data of the participants should not be shared .
Supporting Information: Study Protocol
Time Frame: 3 years

REFERENCES:
- [Result] Langeron O, Birenbaum A, Le Sache F, Raux M. Airway management in obese patient. Minerva Anestesiol. 2014 Mar;80(3):382-92. Epub 2013 Oct 14. PMID 24122033
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/24122033